CLINICAL TRIAL: NCT04962516
Title: Open, Randomized, Parallel Controlled Clinical Trial to Evaluate the Safety and Efficacy of Single-use Precision Filtered Infusion Sets for Intravenous Infusion
Brief Title: Evaluation of the Safety and Efficacy of Single-use Precision Filtered Infusion Sets for Intravenous Infusion
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D2018091
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Single-use Precision Filter Infusion Set
MeSH Terms: interventions — Needles

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group
  Interventions: Device: single-use precision filtered infusion sets
- Control group
  Interventions: Device: single-use precision filter infusion set with needle

INTERVENTIONS:
Device: single-use precision filtered infusion sets — single-use precision filter infusion set (Dalian JMS Medical Apparatus Co., Ltd.)
  Groups: Test group
Device: single-use precision filter infusion set with needle — single-use precision filter infusion set with needle (Shandong Zhongbao Kang Medical Apparatus Co., Ltd.)
  Groups: Control group

SUMMARY:
This study is a pre-market clinical trial of a single-use precision filter infusion set for pumps, to evaluate the safety and effectiveness of a single-use precision filter infusion set for pumps after being used in humans, and to provide clinical evidence for the official application of the product in China

DETAILED DESCRIPTION:
This experiment compares the single-use precision filter infusion set produced by Shandong Xinhua Ande Medical Products Co., Ltd. for the same intended use that has been approved to market, and compares the performance of the two products in clinical use, the overall pass rate, and the occurrence of phlebitis Rates and adverse events are used to evaluate the safety and effectiveness of single-use precision filtration infusion sets for pumps.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older, gender not limited;
2. intravenous infusion requiring drug filtration, flow regulation, dosing and extension of infusion line;
3. not participating in other clinical trials within one month;
4. able to understand the purpose of the trial, voluntarily participate and sign the informed consent;
5. willing to follow up and evaluate according to the requirements of the trial protocol.

Exclusion Criteria:

1. Patients with positive pregnancy test in women of childbearing age or lactating women;
2. Patients with uncontrollable cardiomyopathy, heart failure and unable to tolerate infusion;
3. Patients with uncontrollable decompensated renal function, especially in the anuric phase of acute renal failure and unable to tolerate infusion;
4. Patients with uncontrollable extensive inflammation of the lung parenchyma, pulmonary congestion, pulmonary edema and unable to tolerate infusion;
5. 0.2um size Test devices combined with any of the following drugs or preparations: fatty milk type, blood products type (blood cells, globulin, etc.), drugs that will produce insoluble precipitates with each other, etc.; 6, patients who are clinically infused with very small amounts of drugs (due to residual test line may reduce the amount of drugs delivered to patients); 7, puncture sites with inflammation, tumors, trauma, scars, etc.; 8, those who may be allergic to product materials; 9 Patients with AIDS;

10. Patients with mental disorders; 11. Other patients who are considered by the investigator to be unsuitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Vital signs | 2 hr after injection
  changes in breathing, resting heart rate, blood pressure, body temperature, etc
Vital signs | 24 hr after injection
  changes in breathing, resting heart rate, blood pressure, body temperature, etc
adverse events and complications | 2 hr after injection
  The incidence of adverse events and complications
adverse events and complications | 24 hr after injection
  The incidence of adverse events and complications
number of heat source reactions | 2 hr after injection
  Heat source reactions caused by the application of extension tubes, such as nausea, vomiting, chills, fever, etc., are key safety indicators
number of heat source reactions | 24 hr after injection
  Heat source reactions caused by the application of extension tubes, such as nausea, vomiting, chills, fever, etc., are key safety indicators

CONTACTS AND LOCATIONS:
Overall Officials: Baohua Li, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No